CLINICAL TRIAL: NCT07050602
Title: Long-term Efficacy of Health Belief Model Nursing Intervention in Preventing and Treating Moderate to Severe OSAHS in Post-surgery Patients
Brief Title: Health Belief Model Nursing for Moderate to Severe OSAHS Post-Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, Shuai Chen, Principal investigator, The First Hospital of Hebei Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20160703
Record Dates: First submitted 2025-06-26; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Obstructive Sleep Apnea-Hypopnea Syndrome (OSAHS); Postoperative Care
Keywords: Health Belief Model; Moderate to Severe OSAHS; Postoperative Intervention; Nursing Intervention; Long-term Prevention

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Observation Group (Experimental): Participants received routine postoperative care plus a one-year health belief model nursing intervention. This included: comprehensive assessment and psychological interventions (Perceived Susceptibility); education on OSAHS risks and consequences (Perceived Severity); weekly weight/blood pressure monitoring, dietary/exercise guidance, sleep posture correction aids, and a daily health diary (Perceived Benefits); and regular phone follow-ups (2-3 times/week for 0-8 weeks post-discharge, bi-weekly up to 1 year) for support and addressing difficulties (Perceived Barriers).
  Interventions: Behavioral: Health Belief Model Nursing Intervention; Behavioral: Routine Care
- Control Group (Active Comparator): Participants received routine postoperative care for OSAHS for one year, including general education, dietary and exercise guidance. Post-discharge monitoring was conducted via monthly phone calls.
  Interventions: Behavioral: Routine Care

INTERVENTIONS:
Behavioral: Health Belief Model Nursing Intervention — Participants received a one-year health belief model nursing intervention. This included: comprehensive assessment and psychological interventions (Perceived Susceptibility); education on OSAHS risks and consequences (Perceived Severity); weekly weight/blood pressure monitoring, dietary/exercise guidance, sleep posture correction aids, and a daily health diary (Perceived Benefits); and regular phone follow-ups (2-3 times/week for 0-8 weeks post-discharge, bi-weekly up to 1 year) for support and addressing difficulties (Perceived Barriers).
  Arms: Observation Group
Behavioral: Routine Care — Participants received routine postoperative care for OSAHS for one year, including general education, dietary and exercise guidance. Post-discharge monitoring was conducted via monthly phone calls.

SUMMARY:
This study aimed to investigate the long-term preventive and therapeutic effects of a health belief model (HBM)-based nursing intervention compared to routine care in patients with moderate to severe Obstructive Sleep Apnea-Hypopnea Syndrome (OSAHS) after surgery. The study assessed impacts on sleep parameters (Apnea-Hypopnea Index, Oxygen Desaturation Index, sleep quality via PSQI), self-management abilities, quality of life, OSAHS recurrence rate, and patient satisfaction.

DETAILED DESCRIPTION:
A total of 120 post-surgery patients with moderate to severe OSAHS were recruited and assigned to either a control group (n=60) receiving routine postoperative care or an observation group (n=60) receiving a health belief model-based nursing intervention in addition to routine care. Routine care included general postoperative education for OSAHS, dietary, and exercise guidance with monthly phone follow-ups. The HBM intervention, lasting one year, focused on perceived susceptibility (assessment, psychological intervention), perceived severity (education on risks), perceived benefits (weight/BP monitoring, dietary/exercise guidance, sleep posture aids, daily diary), and perceived barriers (frequent phone follow-ups, psychological support). Outcomes were measured at baseline, 6 months, and 12 months post-surgery, including polysomnography, Pittsburgh Sleep Quality Index (PSQI), self-management ability questionnaires, quality of life questionnaires, OSAHS recurrence, and patient satisfaction surveys.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 30 and 50 years old;
* Sleep Apnea Hypopnea Index (AHI) > 21 events per hour;
* Body Mass Index (BMI) ≥ 28 kg/m²;
* The obstructive plane of OSAHS was either at the soft palate level or associated with narrowing at the tongue base level;
* Surgical treatments included uvulopalatopharyngoplasty (UPPP) or UPPP combined with low-temperature plasma ablation of the tongue base/tongue body;
* The patient had undergone surgical treatment for OSAHS;
* The patient could comprehend the research details and voluntarily signed an informed consent form.

Exclusion Criteria:

* Severe cardiovascular disease, kidney disease, liver disease, or dysfunction of other major organs;
* Severe mental illness or cognitive dysfunction that would hinder understanding or adherence to research procedures;
* Presence of other sleep disorders, such as central sleep apnea or insomnia;
* Use of medications that could interfere with sleep patterns;
* Pregnancy or lactation;
* Patients unwilling to provide informed consent for the study.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Apnea-Hypopnea Index (AHI) | Baseline (immediately after operation) and 6 months post-intervention.
  Measured by Polysomnography (PSG). Lower values indicate better outcome.
OSAHS Recurrence Rate | 6 months and 12 months post-operation.
  Calculated as the percentage of patients experiencing relapse (defined by AHI levels and symptom reappearance) within one year. Lower rates indicate better outcome.

SECONDARY OUTCOMES:
Oxygen Desaturation Index (ODI) | Baseline (immediately after operation) and 6 months post-intervention.
  Measured by Polysomnography (PSG). Lower values indicate better outcome.
Pittsburgh Sleep Quality Index (PSQI) Score | Post-intervention (specific time point after 6 months or 1 year should be clarified, likely at 6 months and/or 1 year).
  Assessed using the PSQI questionnaire (19 questions, 7 components, total score 0-21). Lower scores indicate better sleep quality.
Self-Management Ability | Post-intervention (specific time point, likely at 6 months and/or 1 year).
  Assessed by a questionnaire covering Knowledge Understanding, Adjustment of Daily Life, and Coping Strategies. Each dimension scored 0-10. Higher scores indicate better ability.
Postoperative Quality of Life | Post-intervention (specific time point, likely at 6 months and/or 1 year).
  Assessed by a self-designed questionnaire covering Sleep Quality, Daytime Function, Mental State, and Overall Satisfaction. Each category scored 0-10. Higher scores indicate better quality of life.
Patient Satisfaction with Postoperative Care | 6 months post-intervention.
  Assessed by a survey classifying satisfaction as Very Satisfied, Satisfied, General Satisfaction, Dissatisfied. Total satisfaction rate calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- First Hospital of Hebei Medical University, Shijiazhuang, Hebei, China